CLINICAL TRIAL: NCT00043108
Title: Trimodality Protocol for the Treatment of Locally Advanced, Potentially Resectable Non-Small Cell Lung Cancer Targeting
Brief Title: Combination Chemotherapy, Surgery, and Radiation Therapy in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000256334; P30CA006927 (NIH); NCI-G02-2097 (Other: National Cancer Institutes); 02-014 (Other: FCCC IRB)
Record Dates: First submitted 2002-08-05; First posted 2003-05-07 (Estimated); Results first posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Thoracic RT (50.4 Gy/1.8 Gy Fx) Paclitaxel (50mg/m2/weekly X 6) Carboplatin (AUC 2/weekly X 6)
  Interventions: Drug: carboplatin; Drug: paclitaxel; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving combination chemotherapy with radiation therapy before and after surgery may shrink the tumor so it can be removed during surgery and may kill any remaining tumor cells following surgery.

PURPOSE: Phase II trial to study the effectiveness of combining paclitaxel and carboplatin with radiation therapy and surgery in treating patients who have newly diagnosed locally advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete resection rate and toxic death rate of patients with locally advanced non-small cell lung cancer treated with paclitaxel, carboplatin, and radiotherapy followed by surgical resection and adjuvant paclitaxel and carboplatin.
* Determine the survival, event-free survival, and incidence of pathologic complete remission of patients treated with this regimen.
* Determine the protocol completion rate (CR) of patients treated with this regimen.
* Determine the feasibility and toxicity of this regimen in these patients.
* Determine the pathologic response rate/downstaging, pathologic near CR rate, freedom from distant metastasis rate, and freedom from local regional failure rate of patients treated with this regimen.

OUTLINE: Patients receive induction therapy comprising radiotherapy 5 days a week for 5.5-6 weeks and paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36.

Within 1-3 weeks after completion of induction therapy, patients undergo restaging. Patients with resectable disease undergo surgical resection within 4-8 weeks after induction therapy. Patients with unresectable disease undergo additional radiotherapy 5 days a week for 3 weeks and receive paclitaxel and carboplatin as in induction therapy on days 1, 8, and 15.

Within 4-12 weeks after surgery or additional chemoradiotherapy, patients receive adjuvant therapy comprising paclitaxel and carboplatin as in induction therapy on day 1. Adjuvant treatment repeats every 4 weeks for 3 courses.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 57 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed, newly diagnosed, unilateral primary non-small cell lung cancer (NSCLC)

  * Must have involvement of the superior sulcus, chest wall, or mediastinum
* Must have at least 1 of the following:

  * Locally advanced Pancoast tumors with no documented mediastinal or supraclavicular nodal involvement (T3-T4, N0-1)
  * Resectable chest wall disease (T3, N0-1)
  * Marginally resectable T4, N0-1, or NX central NSCLC
  * N2 patients who are potentially resectable after induction chemoradiotherapy
* No evidence of extrathoracic spread to liver, adrenals, brain, or bone
* No evidence of supraclavicular nodes, malignant pleural or pericardial effusions, or distant metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 3 times upper limit of normal

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No superior vena cava syndrome
* No myocardial infarction within the past 6 months
* No active uncontrolled congestive heart failure
* No active uncontrolled arrhythmia within the past 6 months

Pulmonary

* FEV1 at least 800 mL

Other

* No other active invasive malignancy requiring therapy within the past 2 years
* No ongoing need for adjuvant therapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study entry

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior pelvic or thoracic radiotherapy

Surgery

* See Disease Characteristics

Other

* Concurrent beta blockers, digitalis derivatives, or channel-blocking agents allowed provided cardiac conditions are stable

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2002-07; Primary Completion 2016-12 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aruna J. Turaka, MD, Principal Investigator — Fox Chase Cancer Center; Mark Hallman, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Thoracic RT (50.4 Gy/1.8 Gy Fx) Paclitaxel (50mg/m2/weekly X 6) Carboplatin (AUC 2/weekly X 6)
  carboplatin
  paclitaxel
  conventional surgery
  radiation therapy
Period: Overall Study
Arm/Group | Treatment
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 17
  Black or African American | 2
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Toxic Death Rate
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
Participants | NA — The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and/or is not available to be reported.

2. Primary Outcome: Complete Resection Rates
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
Participants | NA — The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and/or is not available to be reported.

3. Secondary Outcome: Survival
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 19
months | NA [NA to NA] — The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and/or is not available to be reported.

4. Secondary Outcome: Event-free Survival
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 19
months | NA [NA to NA] — The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and/or is not available to be reported.

5. Secondary Outcome: Pathologic Complete Remission (pCR)
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
Participants | NA — The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and/or is not available to be reported.

ADVERSE EVENTS:
Time Frame: 5 years
Description: The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and/or is not available to be reported.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 14/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2004-06-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT00043108/Prot_SAP_ICF_000.pdf